CLINICAL TRIAL: NCT07210216
Title: New Diagnostic Paradigms for the Identification of Early Glaucomatous Damage
Brief Title: GLAUcoma Diagnostic and Imaging Analysis (GLAUDIA) Study
Acronym: GLAUDIA
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6441
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma Open-Angle Primary; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to identify early diagnostic markers of glaucomatous damage by combining functional and structural assessments. Patients with primary open-angle glaucoma and ocular hypertension will undergo comprehensive ophthalmological evaluation, including visual field testing and multimodal imaging of the optic nerve and retina. Both retrospective and prospective data will be collected. The main objective is to define new diagnostic paradigms for detecting early glaucomatous changes and to improve the accuracy of current clinical practice in glaucoma management.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 90 years.
* Best-corrected visual acuity ≥ 0.1 LogMAR (≥ 8/10).
* For primary open-angle glaucoma (POAG):
* IOP ≥ 21 mmHg with normal visual field and/or normal optic nerve head/RNFL, or
* Suspicious optic nerve head (excavation), or
* Reproducible glaucomatous visual field defect.
* POAG patients stratified by visual field mean deviation (MD): -3 to -10 dB (S1-S2 Brusini classification).

Exclusion Criteria:

* Best-corrected visual acuity worse than 0.1 LogMAR (< 8/10).
* Ocular surgery in the last 6 months (except uncomplicated cataract extraction).
* Previous vitreoretinal surgery for macular pathologies (e.g., macular pucker, macular hole) or retinal detachment.
* High myopia (> -3 diopters).
* Optic disc anomalies not attributable to glaucoma (tilted disc, papillary drusen, other morphological/functional anomalies).
* Severe motor disability preventing proper positioning for tests.
* Cognitive impairment reducing test reliability.

Ages: 40 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (40-90 years) with primary open-angle glaucoma, ocular hypertension, or healthy controls, recruited at the Glaucoma Unit, Fondazione Policlinico Universitario A. Gemelli IRCCS.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of early glaucomatous damage detected by multimodal imaging | Baseline to 24 months
  Evaluation of structural parameters from OCT and OCTA and functional indices from visual field testing to detect early glaucomatous damage in ocular hypertensive and glaucoma patients.

SECONDARY OUTCOMES:
Correlation between OCT structural parameters and visual field indices | Baseline to 24 months
  Analysis of the association between RNFL/GCC thickness and visual field MD, PSD, and other indices.